CLINICAL TRIAL: NCT06511661
Title: Prognostic Significance of the Uncertain Resection Based on the Extent of Nodal Dissection for Non-small Cell Lung Cancer: A Propensity Score Matching Retrospective Study
Brief Title: Prognostic Significance of the Uncertain Resection in NSCLC
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mu-Zi Yang, Principal Investigator, Sun Yat-sen University
Other Study IDs: B2024-401
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer; Residual; State
Keywords: Non-small cell lung cancer; Lymphadenectomy; R stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- R0 group: Patients with NSCLC who underwent R0 surgery according to the R stage proposed by IASLC.
  Interventions: Procedure: Complete lymphadenectomy
- R(un) group: Patients with NSCLC who underwent R(un) surgery according to the R stage proposed by IASLC.
  Interventions: Procedure: Incomplete lymphadenectomy

INTERVENTIONS:
Procedure: Complete lymphadenectomy — At least 3 N1 stations and 3 N2 stations are examined during surgery, including station 7.
  Groups: R0 group
Procedure: Incomplete lymphadenectomy — Less than 3 N1 stations or 3 N2 stations are examined during surgery, or those without station 7 lymph node dissection.
  Groups: R(un) group

SUMMARY:
The concept of residual tumor classification proposed by the Union for International Cancer Control (UICC) was used to assess the completeness of surgical resection, and non-small cell lung cancer (NSCLC) patients with incomplete resection were more likely to occur recurrence, leading to significantly poor survival. But this R classification only refers to the surgical margin and neglects other factors associated with surgical quality, such as the extent of lymph node dissection (LND). Therefore, the International Association for the Study of Lung Cancer (IASLC) proposed the definition of uncertain resection [R(un)], which includes the suboptimal extent of LND. However, the clinical significance of R(un) is still controversial. On the one hand, some researches demonstrated that R(un) had definite prognostic significance, with R(un) survival stratifying between R0 and R1. On the other hand, some studies indicated that in early-stage NSCLC, the suboptimal extent of LND had no impact on survival, and the concept of R(un) might be insignificant in these patients. Even in those studies supporting the prognostic significance of R(un), which kind of patients is suitable for R(un) was still unclear. Thus, the investigators explore the impact of the R(un) on the long-term survival of patients with NSCLC using a large cohort in China, to identify those patients who could really benefit from the LND required by the R0 classification proposed by IASLC.

ELIGIBILITY:
Inclusion Criteria:

1. Primary non-small cell lung cancer
2. With pulmonary resection

Exclusion Criteria:

1. Sublobar resection
2. R1/R2
3. Positive highest mediastinal lymph nodes
4. Operative death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data of included patients is extracted from the Hospital Information System of Sun Yat-sen University Cancer Center from 2001 to 2024.
Sampling Method: Non-Probability Sample
Enrollment: 3783 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival | 5 years after surgery
  The disease-free survival rate 5 years after surgery
5-year overall survival | 5 years after surgery
  The overall survival rate 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Zi Yang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China